CLINICAL TRIAL: NCT05534386
Title: How to Prevent Lost in Transition? - Adaptive Randomised Controlled Trial of a Self-management Based Survivorship Intervention for Chinese Cancer Survivors
Brief Title: A Self-management Based Survivorship Intervention for Chinese Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wendy Wing Tak Lam, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW20-100
Record Dates: First submitted 2022-08-31; First posted 2022-09-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Physical Symptom Distress; Weight Management; Neoplasms
Keywords: Physical symptom distress; Weight management; Self-efficacy in managing cancer; Health-related quality of life; Survivorship intervention; Sequential multiple assessment randomized controlled trial; psychooncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: First stage intervention: We will use a block randomization with randomly permuted block sizes of 2,4, and 6 to ensure close balance of the numbers in each arm. Participants will be randomised to the intervention group (i.e. Cancer survivorship care intervention) or control group (i.e. a set of pamphlets explaining symptoms and describing skill-based self-management for symptom management and lifestyle recommendations).
  Second stage intervention: We will use a block randomization with randomly permuted block sizes of 2,4, and 6 to ensure close balance of the numbers in each arm. Participants will be randomised to continue in the trial as usual (i.e. those in the survivorship clinic arm will be asked to follow the advice given by the multidisciplinary team in the initial visit and for those in the control arm will be asked to follow the advices printed in the skill-based self-management pamphlets) or to attend a step-up targeted personalized intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, care provider, investigator and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to intervention or control arms.
  The participants are masked in terms of not knowing that one intervention is hypothesized to yield larger effects than the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- First stage intervention: Cancer survivorship care intervention (CSCI) (Experimental): Patients randomized to the CSCI will attend a 120-minutes survivorship clinic in which each participant will be assessed by members a multidisciplinary team comprising a registered nurse, a dietitian, an exercise physiologist and a psychologist/counsellor. During the visit, participants will receive a personalized (1) treatment summary, (2) assessment and recommendation on managing physical and psychological symptoms, (3) assessment and recommendation on dietary advice, (4) assessment and recommendation on physical activity, and (5) advice on managing potential psychosocial issues. While this is a multidisciplinary clinic, the nurse will be the core facilitator who will give a summary of health assessment report including personalized healthy lifestyle advice and action plan to each participant at the end of the visit.
  Interventions: Behavioral: Cancer survivorship care intervention
- First stage intervention: Control intervention (Active Comparator): Patients randomized to the control group will be given a set of pamphlets explaining symptoms and describing skill-based self-management for symptom management and lifestyle recommendations. Each pamphlet addresses one of the 7 most commonly-reported symptoms (sleep difficulties, fatigue, neuropathy, pain, anxiety, depression, and fear of cancer recurrence) observed in Hong Kong cancer survivors, plus two on lifestyle recommendations (physical activity and healthy diet). All pamphlets are developed based on the self-management framework.
  Interventions: Behavioral: First stage control intervention
- Second stage intervention: Step-up targeted personalized intervention (Experimental): The step-up targeted personalized intervention will adopt a multi-disciplinary approach but place more emphasis on coaching to enhance patient' skills to manage their symptom burden and weight control.
  Interventions: Behavioral: Step-up targeted personalized intervention
- Second stage intervention: Control intervention (Active Comparator): Patients randomized to the control arm at the re-assessment at 4-months post-baseline will continue in the trial as usual (i.e. those in the survivorship clinic arm will be asked to follow the advice given by the multidisciplinary team in the initial visit and for those in the control arm will be asked to follow the advices printed in the skill-based self-management pamphlets).
  Interventions: Behavioral: Second stage control intervention

INTERVENTIONS:
Behavioral: Cancer survivorship care intervention — A one-off face-to-face assessment and personal advice by members of a multidisciplinary team
  Arms: First stage intervention: Cancer survivorship care intervention (CSCI)
Behavioral: Step-up targeted personalized intervention — To provide a more personalized intervention to the participants, but focusing more on symptom management and weight control.
  Arms: Second stage intervention: Step-up targeted personalized intervention
Behavioral: First stage control intervention — A set of skill-based pamphlets will be given.
  Arms: First stage intervention: Control intervention
Behavioral: Second stage control intervention — Those in the survivorship clinic arm will be asked to follow the advice given by the multidisciplinary team in the initial visit and for those in the control arm will be asked to follow the advices printed in the skill-based self-management pamphlet
  Arms: Second stage intervention: Control intervention

SUMMARY:
This study, using a sequential multiple assessment randomized controlled trial (SMART) approach, will evaluate a cancer survivorship care intervention on physical symptom distress, weight management, self-efficacy in managing cancer and health-related quality of life among Chinese patients recently completed curative cancer treatment.

DETAILED DESCRIPTION:
This study, using this SMART approach, will assess the effect of a cancer survivorship care intervention on physical symptom distress, self-efficacy in managing cancer, weight management and health-related quality of life among Chinese patients recently completing curative cancer treatment. First, the investigators will test the effect of a one-off, multidisciplinary team face-to-face assessment (namely, the cancer survivorship clinic) with personalized advice on symptom management, lifestyle modification and anxiety management in reducing the case prevalence of symptom distress, increasing the proportion meeting the weight management criteria, and improving self-efficacy and health-related quality of life among cancer survivors in post-treatment survivorship, in comparison to those receiving skills-based pamphlets for symptom management and lifestyle recommendations. Secondly, this study aims to explore if a step-up targeted personalized intervention is more effective for patients who continue to have symptom distress and/or not to meet the weight management criteria if patients have attended cancer survivorship clinic (i.e. the embedded adaptive intervention) in comparison to those receiving skills-based pamphlets.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese- or Mandarin-speaking Chinese patients diagnosed curable cancer
* have completed primary and adjuvant treatment within the past six months

Exclusion Criteria:

* Patients diagnosed with metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of symptom distress caseness (distress prevalence) | 4-months post-baseline
  The 13-items Edmonton Symptom Checklist (ESAS) will be used to assess symptom distress. The ESAS assesses 13 common symptoms, including pain, fatigue, sleep difficulties, numbness, worrying, feeling sad, or feeling nervous, using a 10-point Likert scale. Patients rating at least one symptom at =>7 will be categorized as moderate-to-severe symptom distress cases.
Proportion of patients with suboptimal weight control | 4-months post-baseline
  Anthropometric measures include weight, height, and body composition, which will be measured in light clothing and without shoes. Weight and body composition including body fat, total body water, muscle mass, bone mass and BMI will be measured using a high-quality segmental body composition monitor (Tanita InnerScan BC545N). Height will be measured to 0.01cm using a portable calibrated stadiometer (SECA Stadiometer). To minimise measurement error, weight and height will be measured twice with accepted values within 0.1kg and 0.3cm, respectively. If either measure falls outside the accepted range, a third measure will be taken. The average of the two acceptable measures will be used in the analysis.
Change in total score of health-related quality of life | Baseline and 4-months post-baseline
  The Standard Chinese version of the European Organization Research Treatment Cancer (EORTC) general quality of life questionnaire (QLQ-C30) will assess health-related quality of life. The EORTC QLQ-C30 includes 30 items that measure five function scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health QoL subscale, five single symptom items (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and financial difficulty.

SECONDARY OUTCOMES:
Change in total scores of self-efficacy | Baseline, 4-months post-baseline, and 12 months post-baseline
  The process outcome is change in total scores of self-efficacy assessed by Self-Efficacy for Managing Chronic Disease scale (SEMCDS) from baseline to 4-months post-baseline, and baseline to 12 months post-baseline. This is a 6-item scale assessing patients' confidence to perform six self-management behaviours. Each item is rated on a 10-point Likert scale. A high score indicates high self-efficacy.
Fear of cancer recurrence | Baseline, 4-months post-baseline, and 12 months post-baseline
  The 42-items Fear of cancer recurrence inventory comprised of seven subscales will be used to assess the change of fear of cancer recurrence (FCR). Each item is rated on a 5-point Likert Scale with a total score ranging from 0 to 168. Higher scores indicate greater FCR. The subscale, Severity will be used as a screening tool for high level of FCR. A score of 13 or higher was optimal for screening.
Illness perception | Baseline, 4-months post-baseline, and 12 months post-baseline
  Cognitive and emotional representations of illness were measured using the nine-item Brief Illness Perception Questionnaire (B-IPQ).
Proportion of symptom distress caseness (distress prevalence) | 12-months post-baseline
  The 13-items Edmonton Symptom Checklist (ESAS) will be used to assess symptom distress. The ESAS assesses 13 common symptoms, including pain, fatigue, sleep difficulties, numbness, worrying, feeling sad, or feeling nervous, using a 10-point Likert scale. Patients rating at least one symptom at =>7 will be categorized as moderate-to-severe symptom distress cases.
Proportion of patients with suboptimal weight control | 12-months post-baseline
  Anthropometric measures include weight, height, and body composition, which will be measured in light clothing and without shoes. Weight and body composition including body fat, total body water, muscle mass, bone mass and BMI will be measured using a high-quality segmental body composition monitor (Tanita InnerScan BC545N). Height will be measured to 0.01cm using a portable calibrated stadiometer (SECA Stadiometer). To minimise measurement error, weight and height will be measured twice with accepted values within 0.1kg and 0.3cm, respectively. If either measure falls outside the accepted range, a third measure will be taken. The average of the two acceptable measures will be used in the analysis.
Health state | Baseline, 4-months post-baseline, and 12 months post-baseline
  Health questionnaire (EQ-5D-5L) including five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression will be used to assessed participants' health state. Each dimension has 5 levels from no problems, slight problems, moderate problems, severe problems to extreme problems. The EQ-5D-5L also records participants self-rated health on a vertical visual analogue scale, where higher values indicate better health the participants can imagine.

OTHER OUTCOMES:
Demographic data | Baseline
  Demographic data including age, gender, marital status, education level, occupation and monthly family income will be assessed by self-reported questionnaire.
Clinical data | Baseline, 4-months post-baseline, and 12 months post-baseline
  Clinical data will be extracted from medical records.
Lifestyle behavior | Baseline, 4-months post-baseline, and 12 months post-baseline
  Lifestyle behavior e.g. drinking and smoking habit will be assessed using a single item question.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wing Tak Lam, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (7):
- Hong Kong (7):
  - Kwong Wah Hospital-Breast Center, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital-Department of oncology, Hong Kong
  - Prince of Wales Hospital-Department of Surgery, Hong Kong
  - Queen Mary Hospital-Department of Obstetrics & Gynaecology, Hong Kong
  - Queen Mary Hospital-Department of Oncology, Hong Kong
  - Queen Mary Hospital-Department of Surgery, Hong Kong
  - Tung Wah Hospital-Department of Surgery, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.